CLINICAL TRIAL: NCT05390242
Title: Peri-implant Marginal Bone Loss and Implant Failure in Patients With Smoking Habit: a Case Control Study
Brief Title: Peri-implant Marginal Bone Loss and Implant Failure in Patients With Smoking Habit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Lina Dumanova, Principal Investigator, University of Barcelona
Other Study IDs: UBMarginalBoneLossStudy
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Dental Implant Failed; Marginal Bone Loss; Smoking
Keywords: Dental Implant
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking Patients with Dental Implantes: Smoking Patients rehabilitated with dental implants at the Dentistry Hospital of the University of Barcelona (Campus of Bellvitge).
  Interventions: Diagnostic Test: Radiographic study
- Non-Smoking Patients with Dental Implantes: Non-Smoking Patients rehabilitated with dental implants at the Dentistry Hospital of the University of Barcelona (Campus of Bellvitge).
  Interventions: Diagnostic Test: Radiographic study

INTERVENTIONS:
Diagnostic Test: Radiographic study — Candidates undergo a radiographic study (Orthopantomography and Implant periapical radiography)

SUMMARY:
The impact of smoking on dental implant failure has been a constant topic of discussion for the past decade and the current literature confronts the inconclusive evidence of tobacco for a marginal bone loss risk factor. The aim of the present investigation is to determine the association between tobacco and marginal bone loss or implant failure in a sample of patients who had received implant-supported restorative therapy in the Dentistry Hospital of the University of Barcelona (Campus of Bellvitge).

Considering that peri-implant marginal bone is essential for dental implant success, in this study we would like to establish the relationship between marginal bone loss around implants and smoking, in our own population study, in order to improve the prognosis of implant success in smoking patients.

On the other hand, knowing the negative effect tobacco has on marginal bone loss in dental implants, we will be able to better predict peri-implant bone loss and reveal the probability of implant failure in short and long-term in smokers. By informing the patient correctly, we can raise awareness and create an additional reason for them to stop smoking, or at least reduce the number of cigarettes they smoke per day.

DETAILED DESCRIPTION:
The present study was designed as a retrospective case control study in a sample of patients with implant-supported restorative therapy conducted at the Dentistry Hospital of the University of Barcelona (Campus of Bellvitge). It is designed following the principles outlined in the Declaration of Helsinki (revised, amended, and clarified in 2013). All of the patients are being properly informed about the study according to the Comité Ético (CEIC) del Hospital Odontològic Universitat de Barcelona guidelines, and informed consent must be signed prior to the interventions. Patients provided with implant-supported restorative therapy were selected from the DHUB database. The sample is divided in two groups: smoking and non-smoking patients. An initial questionnaire is being conducted to obtain information regarding smoking habits. Candidates undergo an oral examination, radiographic study (Orthopantomography and Implant periapical radiograph) and implant probing to determine their peri-implant status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a Smoking Habit
2. Patients 20 - 80 years old
3. Patients rehabilitated at DHUB
4. Patients with a radiographic record at the time of implant loading
5. Patients rehabilitated with one or more dental implants

Exclusion Criteria:

1. Patients with untreated periodontal disease
2. Patients with uncontrolled systemic pathology
3. Pregnant women or in lactation
4. Patients treated with antiresorptive drugs
5. Patients without radiographic records

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients provided with implant-supported restorative therapy selected from the Dentistry Hospital of the University of Barcelona database.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-06-05 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss measured on Periapical Radiography | 60 minutes
  Marginal bone loss (MBL) around dental implants

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontologico de Bellvitge, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar A, Nasreen S, Bandgar S, Bhowmick D, Vatsa R, Priyadarshni P. Comparative Evaluation of Marginal Bone Loss and Implant Failure Rate in Smokers and Nonsmokers. J Pharm Bioallied Sci. 2021 Jun;13(Suppl 1):S203-S206. doi: 10.4103/jpbs.JPBS_676_20. Epub 2021 Jun 5. PMID 34447076
- [Background] Naseri R, Yaghini J, Feizi A. Levels of smoking and dental implants failure: A systematic review and meta-analysis. J Clin Periodontol. 2020 Apr;47(4):518-528. doi: 10.1111/jcpe.13257. Epub 2020 Feb 7. PMID 31955453
- [Background] Linkevicius T, Linkevicius R, Gineviciute E, Alkimavicius J, Mazeikiene A, Linkeviciene L. The influence of new immediate tissue level abutment on crestal bone stability of subcrestally placed implants: A 1-year randomized controlled clinical trial. Clin Implant Dent Relat Res. 2021 Apr;23(2):259-269. doi: 10.1111/cid.12979. Epub 2021 Feb 2. PMID 33527729
- [Background] Nazeer J, Singh R, Suri P, Mouneshkumar CD, Bhardwaj S, Iqubal MA, Dinesh. Evaluation of marginal bone loss around dental implants in cigarette smokers and nonsmokers. A comparative study. J Family Med Prim Care. 2020 Feb 28;9(2):729-734. doi: 10.4103/jfmpc.jfmpc_1023_19. eCollection 2020 Feb. PMID 32318410
- [Background] Badenes-Catalan J, Pallares-Sabater A. Influence of Smoking on Dental Implant Osseointegration: A Radiofrequency Analysis of 194 Implants. J Oral Implantol. 2021 Apr 1;47(2):110-117. doi: 10.1563/aaid-joi-D-19-00223. PMID 32699886
- [Background] Raes S, Rocci A, Raes F, Cooper L, De Bruyn H, Cosyn J. A prospective cohort study on the impact of smoking on soft tissue alterations around single implants. Clin Oral Implants Res. 2015 Sep;26(9):1086-90. doi: 10.1111/clr.12405. Epub 2014 May 5. PMID 24798293
- [Background] Mumcu E, Beklen A. The effect of smoking on the marginal bone loss around implant-supported prostheses. Tob Induc Dis. 2019 May 20;17:43. doi: 10.18332/tid/109279. eCollection 2019. PMID 31516486
- [Background] Javed F, Rahman I, Romanos GE. Tobacco-product usage as a risk factor for dental implants. Periodontol 2000. 2019 Oct;81(1):48-56. doi: 10.1111/prd.12282. PMID 31407428
- [Background] Keenan JR, Veitz-Keenan A. The impact of smoking on failure rates, postoperative infection and marginal bone loss of dental implants. Evid Based Dent. 2016 Mar;17(1):4-5. doi: 10.1038/sj.ebd.6401144. PMID 27012564